CLINICAL TRIAL: NCT02146638
Title: Post Operative Pain Control: Continuous Infusion of Morphine vs Fentanyl. Clinical Outcomes
Brief Title: Post Operative Pain Control: Morphine vs Fentanyl
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Francesca Bevilacqua, medical doctor, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MFN-6932-AS
Record Dates: First submitted 2013-01-10; First posted 2014-05-26 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Post Operative Analgesia
Keywords: post operative analgesia, morphine, fentanyl
MeSH Terms: interventions — Morphine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Morphine (Active Comparator): Patients received morphine 0.02 mg/Kg/h infused at 2 ml/h for 24 hours. The infusion contained morphine and saline.
  Interventions: Drug: Morphine
- Fentanyl (Experimental): Patients received Fentanyl 0.3 mcg/Kg/h infused at 2 ml/h for 24 hours. The infusion contained morphine and saline.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Morphine
  Arms: Morphine
Drug: Fentanyl
  Other Names: Fentanest
  Arms: Fentanyl

SUMMARY:
Aim of this study is to compare benefits and disadvantages in using continuous infusion of morphine or fentanyl for post operative analgesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 or 2 patients
* undergoing major gynaecological surgery

Exclusion Criteria:

* age > 60 years
* obesity (BMI>30 Kg/m2)
* cardiac and respiratory diseases
* renal impairment
* liver disorders
* allergies to any drug used in the study

Ages: 35 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
pain scores | data were recorded during the 24 post operative hours
  data were recorded at 1,6,18 and 24 hours after surgery

SECONDARY OUTCOMES:
analgesic requirements | during the 24 hours after surgery
  if VAS value was equal or higher than 6 patients received ketorolac 30 mg iv

CONTACTS AND LOCATIONS:
Locations (1):
- catholic University of the sacred Heart, Rome, Rome, Italy